CLINICAL TRIAL: NCT01758237
Title: Incidence of Visual Symptom Following Laser (Nd:YAG ) Peripheral Iridotomy (LPI) in Relation to Position of LPI
Brief Title: Dysphotopsia Following Laser Peripheral Iridotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Credit Valley EyeCare (Industry)
Responsible Party: Principal Investigator, Iqbal Ike Ahmed, Principle Investigator, Credit Valley EyeCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVEC-LPI
Record Dates: First submitted 2012-12-20; First posted 2013-01-01 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Narrow Angle Patients at Risk for Angle Closure Glaucoma
Keywords: Laser Peripheral Iridotomy; Visual Dysphotopsia; Visual Disturbances; Angle Closure Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Superior Laser Peripheral Iridotomy (Experimental): Neodymium-doped: Yttrium Aluminum Garnet (Nd:YAG) laser peripheral iridotomy was performed on the superior aspect of the iris in the eye being treated. This will be in the 11 to 1 o'clock position.
  Interventions: Device: Neodymium-doped: Yttrium Aluminum Garnet (Nd:YAG) laser; Procedure: Nd:YAG Laser Peripheral Iridotomy
- Temporal Laser Peripheral Iridotomy (Experimental): Neodymium-doped: Yttrium Aluminum Garnet (Nd:YAG) laser peripheral iridotomy was performed on the temporal aspect of the iris in the eye being treated. The position will be in the 2 to 4 o'clock in the left eye and 8 to 10 o'clock in the right eye.
  Interventions: Device: Neodymium-doped: Yttrium Aluminum Garnet (Nd:YAG) laser; Procedure: Nd:YAG Laser Peripheral Iridotomy

INTERVENTIONS:
Device: Neodymium-doped: Yttrium Aluminum Garnet (Nd:YAG) laser — This device is used to perform the peripheral iridotomy on all patients. It is a standard of care approved device.
  Other Names: Nd:YAG Laser
Procedure: Nd:YAG Laser Peripheral Iridotomy — After application of topical anesthetic to the eye undergoing the LPI, the patient is seated at the laser machine. Abraham iridotomy lens filled with a viscous material will be used to facilitate the procedure. The thinnest area of the iris quadrant treated will be chosen. Nd:YAG Laser will be applied until iridotomy is opened satisfactory.
  Other Names: Nd:YAG LPI

SUMMARY:
To establish the correlation of the location of the Nd:YAG laser peripheral iridotomy to the post operative visual symptoms experienced by some patients. The investigators hypothesize that fully uncovered laser peripheral iridotomy will produce less significant dysphotopsia, due to avoidance of the prismatic effect produced by the tear film than those covered.

DETAILED DESCRIPTION:
Nd:YAG LPI is a frequently performed procedure for patients who have narrow angles at risk of acute angle closure glaucoma, pupillary-block conditions, chronic angle closure, and pigment dispersion syndrome. Most complications associated with the procedure are benign and include intraocular pressure (IOP) spike, transient uveitis, hyphema, corneal or lens damage and closure of the iridotomy. Visual disturbances have been also reported but only a few papers address this specific issue. The rate of these symptoms vary between 2.7% and 4%. It is believed that these symptoms are associated with the fact that light enters through the LPI and thus creating abnormal visual symptoms. Hence it has been suggested to carefully place the LPI so that the eyelid fully covers the LPI, therefore preventing light getting through. However, reports of patients with fully covered LPIs and visual disturbances have led to hypothesize the theory that even when fully covered by the eyelid, light can access through the LPI by a base-up prism created by the tear meniscus at the lid margin. Therefore, placement of the LPI, fully covered, partially covered or totally uncovered can potentially lead to equally significant symptoms. This study will attempt to address the issue of placement of the LPI in relationship with visual symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to make the required study visit
* Able and willing to give consent and follow study instructions
* An indication to undergo laser peripheral iridotomy (narrow angles, occludeable angle at risk of acute angle closure, pupil block condition, chronic angle closure, pigment dispersion syndrome)

Exclusion Criteria:

* Previous intraocular surgery
* Best corrected visual acuity worse than 20/40
* Asymmetrical ptosis of more than 2mm
* Any active intraocular inflammation
* Acute attack of angle closure glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Presence of Linear Dysphotopsia | Baseline (Time =0),1 month
  The change in presence of linear dysphotopsia from baseline (prior to intervention) to 1 month after the Nd:YAG laser intervention is performed.

SECONDARY OUTCOMES:
Presence of Visual Dysphotopsia | Baseline (Time = 0), 1 month
  This includes Halo, Crescent, Ghost Images, Glare, Shadows. This records the change in the presence of these symptoms from baseline (prior to intervention) and 1 month after the Nd:YAG laser intervention.
Pain Experienced | Procedure (Time = 0)
  The pain experienced when the Nd:YAG procedure is performed. This is on a scale of 0-10 with 0 being no pain and 10 the most severe pain imaginable.
Nd:YAG Laser Power Used | Procedure (Time = 0)
  The amount of laser power used on the Nd:YAG laser to perform the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Ike K Ahmed, MD, Principal Investigator — University of Toronto, Toronto, Canada. University of Utah, Salt Lake City, USA; Vanessa Vera, MD, Study Director — University of Toronto, Canada
Locations (1):
- Credit Valley EyeCare, Mississauga, Ontario, Canada

REFERENCES:
- [Background] Khodadoust AA, Arkfeld DF, Caprioli J, Sears ML. Ocular effect of neodymium-YAG laser. Am J Ophthalmol. 1984 Aug 15;98(2):144-52. doi: 10.1016/0002-9394(87)90348-5. PMID 6548087
- [Background] Murphy PH, Trope GE. Monocular blurring. A complication of YAG laser iridotomy. Ophthalmology. 1991 Oct;98(10):1539-42. doi: 10.1016/s0161-6420(91)32091-8. PMID 1961641
- [Background] Spaeth GL, Idowu O, Seligsohn A, Henderer J, Fonatanarosa J, Modi A, Nallamshetty HS, Chieh J, Haim L, Steinmann WC, Moster M. The effects of iridotomy size and position on symptoms following laser peripheral iridotomy. J Glaucoma. 2005 Oct;14(5):364-7. doi: 10.1097/01.ijg.0000177213.31620.02. PMID 16148584
- [Background] Weintraub J, Berke SJ. Blurring after iridotomy. Ophthalmology. 1992 Apr;99(4):479-80. doi: 10.1016/s0161-6420(92)38516-1. No abstract available. PMID 1584561
- [Background] Congdon N, Yan X, Friedman DS, Foster PJ, van den Berg TJ, Peng M, Gangwani R, He M. Visual symptoms and retinal straylight after laser peripheral iridotomy: the Zhongshan Angle-Closure Prevention Trial. Ophthalmology. 2012 Jul;119(7):1375-82. doi: 10.1016/j.ophtha.2012.01.015. Epub 2012 Mar 14. PMID 22424576
- [Background] Chung RS, Guan AE. Unusual visual disturbance following laser peripheral iridotomy for intermittent angle closure glaucoma. Graefes Arch Clin Exp Ophthalmol. 2006 Apr;244(4):532-3. doi: 10.1007/s00417-005-0129-x. Epub 2005 Oct 14. No abstract available. PMID 16228219
- [Derived] Vera V, Naqi A, Belovay GW, Varma DK, Ahmed II. Dysphotopsia after temporal versus superior laser peripheral iridotomy: a prospective randomized paired eye trial. Am J Ophthalmol. 2014 May;157(5):929-35. doi: 10.1016/j.ajo.2014.02.010. Epub 2014 Feb 14. PMID 24531024